CLINICAL TRIAL: NCT07112898
Title: Effect of Platelet-Rich Plasma on Graft Uptake and Postoperative Outcomes in Full-Thickness Skin Grafting of Face and Neck
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Irfan Jamil, Principal Investigator, Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LahoreGeneralH5
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Skin Transplantation; Reconstructive Surgical Procedures
Keywords: Full-Thickness Skin Graft; Platelet-Rich Plasma; Wound Healing Enhancement; Graft Uptake

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PRP (Experimental): Patients in this group received autologous platelet-rich plasma (PRP) applied to both the recipient wound bed and the graft before graft placement, during full-thickness skin grafting for facial or neck defects.
  Interventions: Procedure: Platelet-Rich Plasma (PRP)
- Group Control (Active Comparator): Patients in this group underwent standard full-thickness skin grafting on the face or neck without PRP application.
  Interventions: Procedure: Standard Skin Grafting

INTERVENTIONS:
Procedure: Platelet-Rich Plasma (PRP) — Autologous PRP (approximately 4-6 mL) will be prepared using a double centrifugation technique and activated with 10% calcium gluconate. It will be administered by injecting 0.1-0.2 mL/cm² subdermally into the recipient bed and intradermally into the graft prior to placement.
  Other Names: Autologous PRP
  Arms: Group PRP
Procedure: Standard Skin Grafting — Grafts will be placed on a clean, vascularized wound bed, secured with nonabsorbable sutures, and covered with standard postoperative dressings. No PRP will be applied.
  Other Names: Conventional Full-Thickness Skin Graft
  Arms: Group Control

SUMMARY:
This clinical study aims to evaluate whether applying platelet-rich plasma (PRP), a substance made from a person's own blood, can improve the success of full-thickness skin grafts used to treat facial and neck wounds. Skin grafting is a common reconstructive technique for covering wounds caused by injuries, burns, surgeries, or other conditions. However, skin grafts sometimes do not heal well, leading to complications such as graft failure, infection, or delayed healing, especially in delicate areas like the face and neck.

Platelet-rich plasma contains special healing components called growth factors that may help tissues heal faster and better. These growth factors support new blood vessel formation, reduce swelling, and promote healthy skin regeneration. In this study, participants will be randomly assigned to one of two groups. One group will receive skin grafts along with PRP applied to the wound and graft site, while the other group will receive standard grafting without PRP.

The study will measure how much of the graft survives and integrates into the wound (called "graft uptake") on the 7th day after surgery. It will also assess other early outcomes such as signs of redness (erythema), infection, or blood collection under the graft (hematoma). The hypothesis is that using PRP will lead to better graft healing and fewer complications than using skin grafts alone. The results of this study may help improve recovery and reduce the need for further procedures in patients with facial and neck skin defects.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years undergoing full-thickness skin grafting for facial or cervical skin defects.
* Indications for grafting include post-traumatic defects, burns, tumor excision, or revision surgeries.
* Patients with wound defects of size ranging between 3 cm² and 6 cm², amenable to single-session full-thickness skin grafting.
* Patients in whom the recipient bed is healthy, vascularized, and free of necrotic tissue at the time of surgery.

Exclusion Criteria:

* Patients with systemic conditions known to impair wound healing, including uncontrolled diabetes mellitus (HbA1c >8%), severe peripheral vascular disease, collagen vascular disorders, or immunodeficiency.
* Patients with hematological disorders affecting platelet count or function, including thrombocytopenia (platelet count <150,000/µL), coagulopathies, or platelet dysfunction syndromes.
* Patients on systemic anticoagulation therapy (e.g., warfarin, DOACs) or corticosteroids within the last 4 weeks.
* Presence of active local infection or purulent discharge at the recipient or donor site at the time of surgery.
* History of previous radiation to the grafted site or underlying malignancy with ongoing treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Graft Uptake at Day 7 Postoperatively | 7th postoperative day
  Graft uptake will be assessed as the percentage of the original wound area successfully covered by the viable graft on the 7th postoperative day. This will be calculated using the formula:
  Graft Uptake (%) = [(Original wound area - Denuded area) ÷ Original wound area] × 100.
  The denuded area will be determined using sterile measurement tools such as a surgical ruler, grid tracing, or digital planimetry. Based on the uptake percentage, the graft will be categorized qualitatively as: Excellent (>90%), Good (76-90%), Moderate (50-75%), Poor (<50%), or Failed (0%).

SECONDARY OUTCOMES:
Proportion of Patients with Graft Failure (0% Uptake) | 7th postoperative day
  Graft failure will be defined as complete necrosis or detachment of the graft, resulting in 0% uptake on the 7th postoperative day. Failure will be confirmed through clinical evaluation and photographic documentation.
Local Graft Site Infection | 7th postoperative day
  Infection will be diagnosed if at least two of the following signs are present: purulent discharge, localized swelling, increased warmth, or breakdown at the graft margins. Evaluation will be performed by the surgical team, and swabs may be collected if purulent discharge is observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore General Hospital, Lahore, Lahore, Punjab Province, Pakistan